CLINICAL TRIAL: NCT04063488
Title: An Observational Study of the Effects of Metreleptin in Young Adults With Congenital Leptin Deficiency
Brief Title: The Effects of Metreleptin in Congenital Leptin Deficiency
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Lisa Neff, Associate Professor, Endocrinology, Metabolism and Molecular Medicine, Northwestern University
Other Study IDs: 00209730
Record Dates: First submitted 2019-07-12; First posted 2019-08-21 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Congenital Leptin Deficiency (Disorder)
MeSH Terms: interventions — metreleptin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Metreleptin — This is an observational study in which the subjects will serve as their own controls. Study testing will be conducted at baseline (pre-treatment) and for 2 years, post-treatment with metreleptin.
  Other Names: Myalept

SUMMARY:
This study has been designed to 1) provide access to metreleptin to the only two individuals in the US known to have congenital leptin deficiency (CLD) and 2) explore a variety of unanswered questions about leptin physiology in general and metreleptin therapy in CLD specifically.

The primary study endpoints include the following measures: body composition, measures of hepatic steatosis, measures of insulin sensitivity, and measures of sleep architecture.

Secondary study endpoints include assessment of clock gene expression, body temperature, thyroid function, gonadal function, cognitive function, eating behavior, physical activity, mood, quality of life, and body image.

DETAILED DESCRIPTION:
Congenital leptin deficiency (CLD) is a rare autosomal recessive condition caused by a mutation in the leptin gene (LEP). This mutation leads to a severe deficiency in leptin, a hormone secreted primarily by adipocytes. Leptin is also secreted by gastric mucosal cells, in response to stimuli such as food intake. Leptin has many important physiologic roles, including serving as a signal to the hypothalamus of both long-term (adipocyte) and short-term (gastric) energy storage. Individuals with CLD have hyperphagia and morbid obesity with an onset in early childhood. Hypogonadotropic hypogonadism, insulin resistance, and immune dysfunction are also often observed in patients with CLD but these features can be of varying degrees of severity.

Recombinant human leptin (metreleptin; Myalept®) was approved by the U.S. Food and Drug Administration in 2014 to treat the complications of leptin deficiency in patients with generalized lipodystrophy (GL). Commercial use of metreleptin is restricted to patients with leptin deficiency due to GL. However, ~3 dozen patients worldwide who are known to have congenital leptin deficiency (CLD) have been treated safely and successfully with metreleptin in the investigational setting for two decades. Metreleptin therapy has been shown to reduce hunger and desire to eat in leptin-deficient humans, and significant weight loss is typical.

Some questions remain regarding the pluripotent effects of metreleptin in patients with CLD. Understudied aspects of physiology in these patients include the role of leptin (independent of weight) in insulin sensitivity, hepatic steatosis, and sleep. For each of these areas, there is preliminary evidence from humans or the ob/ob (leptin-deficient) mouse model for a beneficial role of leptin, but important knowledge gaps remain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital leptin deficiency
* Age 18 years or older
* Must agree to use contraception for the duration of treatment with metreleptin and for 6 months post-treatment completion.

Exclusion Criteria:

* Presence of a clinically significant medical condition that could significantly affect the risk/benefit ratio for metreleptin treatment, as judged by the PI
* Known allergies to E. coli-derived proteins or hypersensitivity to any component of metreleptin treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll two young adults who have been recently diagnosed with congenital leptin deficiency (homozygous for the pathogenic variant c.398delG in exon 3 of the leptin gene). They have not been previously treated with metreleptin.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
change in hepatic steatosis | repeated measures at baseline, 1 week, 1 month, 3 months, 6 months, 12 months, 18 months, 24 months
  ultrasound elastography with dispersion imaging
change in insulin sensitivity | repeated measures at baseline, 1 week, 3 months
  HOMA (fasting labs)
change in sleep architecture | repeated measures at baseline, 3 months, 6 months, 12 months
  polysomnography
change in body composition | repeatured measures at baseline, 3 months, 6 months, 12 months, 18 months, 24 months
  full body DXA

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Neff, MD, Principal Investigator — Dr.
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States